CLINICAL TRIAL: NCT04676295
Title: Pre-eclampsia and Future Cardiovascular Health: An Underused Opportunity to Improve Family Health
Acronym: FINNCARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Tiina Jääskeläinen, Principal Investigator, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FINNCARE
Record Dates: First submitted 2020-12-07; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Pre-Eclampsia; Cardiovascular Diseases; Cardiovascular Risk Factor; Gestational Hypertension
MeSH Terms: conditions — Pre-Eclampsia; Cardiovascular Diseases; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PE intervention (Experimental): A 12-month lifestyle intervention program to improve mothers and their children blood pressure and CVD risk profile.
  Interventions: Behavioral: Face-to-face and web-based lifestyle intervention
- PE control (No Intervention): The control group continue habitual lifestyle but will perform the same baseline and follow-up measurements as the intervention group. They will be given general written information on healthy eating.
- Non-PE control (No Intervention): The control group continue habitual lifestyle but will perform the same baseline and follow-up measurements as the intervention group. They will be given general written information on healthy eating.

INTERVENTIONS:
Behavioral: Face-to-face and web-based lifestyle intervention — Families are provided at baseline with one 60 min face-to-face dietary counseling session with nutritionist using family-oriented motivational interviewing and solution focusing techniques. The intervention continues in an interactive web-based portal where different modules include assignments, activities, and tests and related videos targeting five cardiovascular health-linked behaviors: 1) improving quality of fat in the diet, 2) increasing the consumption of foods rich in fiber, 3) decreasing the use of salt, 4) increasing physical activity and 5) reducing smoking.
  Arms: PE intervention

SUMMARY:
Background: PE (pre-eclampsia) is a common pregnancy-specific vascular hypertensive disease affecting 3-5% of pregnancies. PE independently increases the risk for premature cardiovascular disease (CVD) in mothers and their offspring long-term. PE provides a unique window for early risk profiling and CVD prevention. However, the efficacy of a family oriented lifestyle intervention to lower CVD risk in families with history of PE has not previously been evaluated.

Aim: This study will explore the impact of PE on CVD progression 8-12 years from delivery in mothers and their children, and assess whether a lifestyle intervention is useful for lowering mother and child blood pressure and improving the CVD risk profile overall in families with a history of PE.

Hypothesis: PE is related with CVD progression mediated by elevated blood pressure. Blood pressure and the CVD risk profile overall is modifiable in mothers and children by a 12-month behavioral lifestyle intervention in families with a history of PE.

Study design: Randomized controlled behavioral lifestyle intervention trial where families (mother, child and father from the FINNPEC study) are offered the opportunity to participate in a lifestyle intervention program 8-12 years after a PE pregnancy. 300 PE families will be randomized 1:1 to a 12-month lifestyle intervention program or to a control group. A parallel group of 100 non-PE control families will be assessed at baseline and follow-up.

Main outcome: 24 hour mean blood pressure change between baseline and follow-up in mother and child.

Significance: This study will provide information on CVD progression in mothers and children 8-12 years from a PE pregnancy. Furthermore, the study assess the effect of a 12-month lifestyle intervention on blood pressure and CVD risk profile overall following a PE pregnancy. Potentially, the study provides the opportunity to identify PE families at highest risk of CVD progression and families amenable to blood pressure and CVD risk profile improvement.

DETAILED DESCRIPTION:
Power analysis:

Power calculations were performed in order to detect 5.5 mmHg reduction in maternal systolic blood pressure with a power of 80% and a 2-sided p-value of 0.05 for the difference between the groups (intervention and control PE) (NICE 2011). Accounting for a 20% loss to follow-up or missing data, a sample of 148 women in the PE intervention group and 148 women in the PE control group is needed.

Specific objectives:

1. To assess cardiovascular health and CVD progression in families (mother, child and father) 8-12 years following a PE pregnancy compared with non-PE control families.
2. To assess the effectiveness of a behavioral 12-month lifestyle intervention in mothers and their children 8-12 years following a PE pregnancy to lower blood pressure and improve their CVD risk profile overall.
3. To assess the effectiveness of a lifestyle intervention on the awareness of CVD risk after a PE pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Families are recruited from the FINNPEC cohort. In FINNPEC, PE was defined as hypertension and proteinuria occurring after 20 weeks gestation (American College of Obstetricians and Gynecologists 2002 criteria). Hypertension was defined as systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg. Proteinuria was defined as urinary excretion of ≥0.3 g protein in a 24-hour specimen, or 0.3 g/L, or two ≥1+ readings on a dipstick in a random urine determination with no evidence of a urinary tract infection. Each PE diagnosis was ascertained based on hospital records and confirmed independently by a research nurse and a study physician in the original FINNPEC case-control study including 1450 nulliparous or multiparous women with a singleton pregnancy with PE and 1065 pregnant control women without PE (aged 18-47 years) from all 5 university hospitals in Finland during 2008-2011.

Exclusion criteria in the FINNPEC: multiple pregnancy, inability to speak Finnish or Swedish.

Exclusion Criteria in the FINNCARE:

* Pregnancy and/or lactation (for all mothers)
* Pre-eclampsia in any previous or subsequent pregnancies (for all non-PE mothers)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure (mothers) | baseline -12 months
  mean 24 hour ambulatory systolic BP and diastolic BP; mmHg
Blood pressure (children) | baseline -12 months
  mean 24 hour ambulatory systolic BP and diastolic BP; mmHg

SECONDARY OUTCOMES:
Blood pressure 24 hour variability (mothers) | baseline -12 months
  nocturnal systolic and diastolic BP dip; standard deviation of systolic and diastolic BP; weighted standard deviation of systolic and diastolic BP; mmHg
Arterial stiffness (mothers) | baseline -12 months
  carotid-femoral pulse wave velocity; m/s
Adiposity (mothers) | baseline -12 months
  BMI; kg/m2
Adiposity (mothers) | baseline -12 months
  waist-hip-ratio (no unit)
Adiposity (mothers) | baseline -12 months
  body fat percentage; %
Dietary intake (mothers) | baseline -12 months
  food frequency questionnaire on quality of fat (SFA, MUFA and PUFA; E%/day)
Dietary intake (mothers) | baseline -12 months
  food frequency questionnaire on fiber intake; g/day
Dietary intake (mothers) | baseline -12 months
  food frequency questionnaire on salt intake; g/d
Physical activity and sedentary behavior (mothers) | baseline -12 months
  questionnaire data: weekly number of sessions and minutes of moderate-to-vigorous-intensity physical activity and walking
Physical activity and sedentary behavior (mothers) | baseline -12 months
  questionnaire data: meeting physical activity recommendations
Physical activity and sedentary behavior (mothers) | baseline -12 months
  questionnaire data: daily minutes of sitting on a non-weekend and weekend day
Physical activity and sedentary behavior (mothers) | baseline -12 months
  accelerometer data: daily number of steps
Physical activity and sedentary behavior (mothers) | baseline -12 months
  accelerometer data: daily minutes of total and intensity-specific physical activity
Physical activity and sedentary behavior (mothers) | baseline -12 months
  accelerometer data: daily minutes of stationary behavior
Physical activity and sedentary behavior (mothers) | baseline -12 months
  accelerometer data: daily number of breaks in stationary behavior
Smoking (mothers) | baseline -12 months
  questionnaire on status of smoking/use of snuf/use of electronic cigarettes/nicotine replacement therapy and number of cigarettes/day
Laboratory assessment of cardiovascular risk (mothers) | baseline -12 months
  lipids (total cholesterol, LDL, HDL, triglycerides; mmol/l)
Laboratory assessment of cardiovascular risk (mothers) | baseline -12 months
  hs-CRP; mg/l
Laboratory assessment of cardiovascular risk (mothers) | baseline -12 months
  HOMA index calculated as glucose; mmol/l x insulin; mU/l / 22.5
Awareness of later life morbidity (mothers) | baseline -12 months
  A brief questionnaire with true or false questions on pre-eclampsia and later life morbidity
Heart rate variability (mothers) | baseline -12 months
  standard deviation of all R-R intervals; root mean square of successive R-R interval differences, ms; High frequency power of R-R intervals from spectral band 0.15-0.4 Hz, ms2 ;Low frequency power of R-R intervals from spectral band 0.04-0.15 Hz, ms2 ; and LF/HF ratio
Blood pressure 24 hour variability (children) | baseline -12 months
  nocturnal systolic and diastolic BP dip; standard deviation of systolic and diastolic BP; weighted standard deviation of systolic and diastolic BP; mmHg
Arterial stiffness (children) | baseline -12 months
  carotid-femoral pulse wave velocity; m/s
Adiposity (children) | baseline -12 months
  BMI z-score
Adiposity (children) | baseline -12 months
  waist-hip-ratio (no unit)
Adiposity (children) | baseline -12 months
  body fat percentage; %
Dietary intake (children) | baseline -12 months
  food frequency questionnaire derived data on SFA index, fiber index, salt index (sum of food items rich in SFA/fiber/salt used during the previous week)
Physical activity and sedentary behavior (children) | baseline -12 months
  questionnaire data: weekly number of days and daily duration of active travel to school and hobbies, structured physical activity outside school hours, unstructured physical activity outside school hours, screen time sitting, non-screen time sitting Accelerometer data: daily number of steps; daily minutes of total and intensity-specific physical activity; daily minutes of and stationary behavior; meeting physical activity recommendations; daily number of breaks in stationary behavior
Physical activity and sedentary behavior (children) | baseline -12 months
  questionnaire data: weekly number of days and daily duration of active travel to school and hobbies
Physical activity and sedentary behavior (children) | baseline -12 months
  questionnaire data: structured physical activity outside school hours
Physical activity and sedentary behavior (children) | baseline -12 months
  questionnaire data: unstructured physical activity outside school hours
Physical activity and sedentary behavior (children) | baseline -12 months
  questionnaire data: screen time and non-screen time sitting
Physical activity and sedentary behavior (children) | baseline -12 months
  accelerometer data: daily number of steps
Physical activity and sedentary behavior (children) | baseline -12 months
  accelerometer data: daily minutes of total and intensity-specific physical activity
Physical activity and sedentary behavior (children) | baseline -12 months
  accelerometer data: daily minutes of stationary behavior
Physical activity and sedentary behavior (children) | baseline -12 months
  accelerometer data: meeting physical activity recommendations
Physical activity and sedentary behavior (children) | baseline -12 months
  accelerometer data: daily number of breaks in stationary behavior
Laboratory assessment of cardiovascular risk (children) | baseline -12 months
  lipids (total cholesterol, LDL, HDL, triglycerides; mmol/l)
Laboratory assessment of cardiovascular risk (children) | baseline -12 months
  hs-CRP; mg/l
Laboratory assessment of cardiovascular risk (children) | baseline -12 months
  HOMA index calculated as glucose; mmol/l x insulin; mU/l / 22.5
Process evaluation: reach | baseline
  participation rate of the families recruited (research database on study visits)
Process evaluation: reach | baseline
  representativeness of the families participating (parents' and children's age, questionnaire on socio-economics)
Process evaluation: compliance | baseline -12 months
  participation rate in measurements (number of study visits and questionnaires completed)
Process evaluation: compliance | baseline -12 months
  proportion of sessions completed in the web-based portal (data accumulated in the web-based portal)
Process evaluation: acceptability | baseline -12 months
  usefulness and ease of use (questionnaire and proportion of webportal sessions completed by the families)
Process evaluation: acceptability | baseline -12 months
  credibility and satisfaction of the web-based portal (questionnaire and proportion of webportal sessions completed by the families)
Process evaluation: acceptability | baseline -12 months
  occurrence of technical problems (questionnaire)

OTHER OUTCOMES:
Arterial wall thickness (mothers) | baseline
  intima-media thickness; common carotid, brachial and radial; mm
Left ventricular mass (mothers) | baseline
  left ventricular mass; g
Left ventricular systolic function (mothers) | baseline
  left ventricular global longitudinal strain; %
Left ventricular diastolic function (mothers) | baseline
  left atrial volume; ml
Left ventricular diastolic function (mothers) | baseline
  pulsed wave Doppler mitral early to late inflow velocity ratio (no unit)
Left ventricular diastolic function (mothers) | baseline
  mitral lateral annular pulsed wave tissue Doppler early velocity; cm/s
Left ventricular diastolic function (mothers) | baseline
  septal pulsed wave tissue Doppler early velocity; cm/s
Arterial wall thickness (children) | baseline
  intima-media thickness; common carotid, brachial and radial; mm
Left ventricular mass (children) | baseline
  left ventricular mass; g
Left ventricular systolic function (children) | baseline
  left ventricular global longitudinal strain; %
Left ventricular diastolic function (children) | baseline
  left atrial volume; ml
Left ventricular diastolic function (children) | baseline
  pulsed wave Doppler mitral early to late inflow velocity ratio (no unit)
Left ventricular diastolic function (children) | baseline
  mitral lateral annular pulsed wave tissue Doppler early velocity; cm/s
Left ventricular diastolic function (children) | baseline
  septal pulsed wave tissue Doppler early velocity; cm/s

CONTACTS AND LOCATIONS:
Overall Officials: Tiina Jääskeläinen, PhD, Principal Investigator — University of Helsinki; Hannele Laivuori, Prof, MD, Study Chair — University of Helsinki and University of Tampere; Taisto Sarkola, PhD, MD, Study Director — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

REFERENCES:
- [Result] Jaaskelainen T, Heinonen S, Kajantie E, Kere J, Kivinen K, Pouta A, Laivuori H; FINNPEC Study Group. Cohort profile: the Finnish Genetics of Pre-eclampsia Consortium (FINNPEC). BMJ Open. 2016 Nov 10;6(11):e013148. doi: 10.1136/bmjopen-2016-013148. PMID 28067621
- [Derived] Renlund-Vikstrom M, Jaaskelainen TJ, Kivela A, Heinonen S, Laivuori H, Sarkola T. Cardiac Structure and Function in 8- to 12-Year-Old Children Following In-Utero Exposure to Preeclampsia (FINNCARE Study). J Am Heart Assoc. 2024 Aug 6;13(15):e034494. doi: 10.1161/JAHA.124.034494. Epub 2024 Jul 16. PMID 39011963
- [Derived] Renlund MA, Jaaskelainen TJ, Kivela ASE, Heinonen ST, Laivuori HM, Sarkola TA. Blood pressure, arterial stiffness, and cardiovascular risk profiles in 8-12-year-old children following preeclampsia (FINNCARE-study). J Hypertens. 2023 Sep 1;41(9):1429-1437. doi: 10.1097/HJH.0000000000003485. Epub 2023 Jun 19. PMID 37337860